CLINICAL TRIAL: NCT05893394
Title: Core Stability as a Prognostic Factor of Urinary Incontinence in Patients Undergoing Robot-assisted Laparoscopic Prostatectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: CLF 23/01
Record Dates: First submitted 2023-05-30; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims at investigating the possible correlation between core stability muscles and urinary incontinence following Robot-Assisted Laparoscopic Prostatectomy.

Sixty-two patients who are candidates for Robot-Assisted Laparoscopic Prostatectomy will be enrolled. All participants will be asked to be evaluated in their core stability functionality 30-40 days before Robot-Assisted Laparoscopic Prostatectomy intervention. The core stability functionality result will be correlated with the urinary incontinence 45-50 days after intervention.

DETAILED DESCRIPTION:
The study aims at investigating the correlation between core stability muscles and urinary incontinence following Robot-Assisted Laparoscopic Prostatectomy.

All sixty-two participants will be asked to be evaluated in their core stability functionality 30-40 days before Robot-Assisted Laparoscopic Prostatectomy intervention. Core stability functionality will be evaluated through the Loumajoki Battery of tests, composed of 10 simple items in which the patients have to maintain core stability. In addition a Quality of Life questionnaire (WHO Quality of Life-BREF) will be administered. The core stability functionality result will be correlated with urinary incontinence measured by the 24h PAD test 45-50 days after intervention. At this point core stability will be evaluated again as done before.

ELIGIBILITY:
Inclusion Criteria:

* Patient who are candidates for Robot-Assisted Laparoscopic Prostatectomy
* Objectivity of core muscles recruitment through the Loumajoki Battery

Exclusion Criteria:

* Pre-surgery incontinence
* Pre-intervention radiotherapy treatment
* Previous urogenital surgery
* Concomitant presence of neurological, internal medicine or musculoskeletal system pathologies that may affect functional or motor recovery
* Subjects with cognitive deficits and/or psychiatric disorders
* Lumbar stabilization or abdominal interventions
* Acute low back pain

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing Robot-Assisted Laparoscopic Prostatectomy
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between Core stability functionality and Urinary Incontinence. | Core stability evaluated 30-40 days before surgery. Urinary incontinence evaluated 45-50 days after surgery
  To evaluate any correlation between Core stability functionality measured with Loumajoki Battery and Urinary Incontinence measured with 24h PAD test.

SECONDARY OUTCOMES:
Correlation between Core stability functionality and Quality of Life. | Core stability evaluated 30-40 days before surgery. Quality of Life evaluated 30-40 days before surgery
  To evaluate any correlation between Core stability functionality measured with Loumajoki Battery and Quality of Life measured with WHO Quality of Life-BREF.
Variation between Core stability functionality at base line and at follow-up. | Core stability evaluated 30-40 days before surgery and 45-50 days after surgery
  To evaluate any variation between Core stability functionality at base line and at follow-up measured with Loumajoki Battery.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Italy